CLINICAL TRIAL: NCT06015568
Title: Phase I Study of Anti-EGFR/c-Met Bispecific Antibody MCLA-129 Combined With Befotertinib in Patients of Advanced Non-small Cell Lung Cancer With EGFR Sensitive Mutation To Evaluate The Safety, Pharmacokinetic Characteristics and Antitumor Activity
Brief Title: Study of MCLA-129 Combined With Befotertinib in the Treatment of Advanced Non-small Cell Lung Cancer With EGFR Sensitive Mutation
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Betta Pharmaceuticals Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BTP-21712
Record Dates: First submitted 2023-08-21; First posted 2023-08-29 (Actual); Last update posted 2023-08-29 (Actual); Status verified 2023-08

CONDITIONS: Non-Small Cell Lung Cancer、EGFR Sensitive Mutation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- MCLA-129+ Befotertinib (Experimental): Drug:MCLA-129 1500mg or 2000mg IV Q2W Other name:MCLA-129 Drug:Befotertinib (75 mg or 100 mg orally, once daily) Other name:D-0316
  Interventions: Drug: MCLA-129: 1500mg or 2000mg IV Q2W; Drug: Befotertinib: 75 mg or 100 mg Po QD

INTERVENTIONS:
Drug: MCLA-129: 1500mg or 2000mg IV Q2W — Every 28 days is a cycle until disease progression, death, initiation of new anti-tumor treatment, loss of follow-up, or voluntary withdrawal occurs
Drug: Befotertinib: 75 mg or 100 mg Po QD — The initial dose of Befotertinib is 75 mg orally once daily (QD) for one cycle, and then increased to 100 mg orally QD in the absence of CTCAE grade ≥ 2 headache or thrombocytopenia during the first cycle, otherwise maintained to 75 mg orally QD.
  Every 28 days is a cycle until disease progression, death, initiation of new anti-tumor treatment, loss of follow-up, or voluntary withdrawal occurs.

SUMMARY:
To evaluate the safety and tolerance of MCLA-129 combined with Befotertinib in patients with advanced non-small cell lung cancer with EGFR-sensitive mutations.

DETAILED DESCRIPTION:
This is a phase I study to evaluate the safety, pharmacokinetic characteristics and antitumor activity of anti-EGFR/c-Met bispecific antibody MCLA-129(1500mg Q2W IV or 2000mg Q2W IV) combined with Befotertinib (75 mg once daily for first cycle, then increased to 100 mg once daily, orally) in Patients of advanced non-small cell lung cancer with exon 19 deletion or exon 21 L858R mutation(either alone or in combination with other EGFR mutations).

ELIGIBILITY:
Inclusion Criteria:

* Age from 18 to 75 years.
* Histologically or cytologically confirmed locally advanced or metastatic NSCLC that is not suitable for radical surgery or radiotherapy, and harbored EGFR exon 19 deletion or exon 21 L858R mutation( either alone or in combination with other EGFR mutations) in NSCLC assessed by genetic testing.
* For Part 1: patients with advanced NSCLC must be progression, or intolerance, or rejected to standard therapy(subjects treated with Befotertinib must be progression of the disease).
* For Part 2, each cohort is defined as follows:

  * Cohort A: Previously diagnosed EGFR-sensitive mutations and no systemic antitumor therapy for locally advanced or metastatic NSCLC.
  * Cohort B: Advanced NSCLC patients with previously diagnosed EGFR-sensitive mutations and third generation EGFR-TKI resistance.
  * Cohort C: Advanced NSCLC patients who had previously been diagnosed with EGFR-sensitive mutations and first or second EGFR-TKI resistance.

Patients in cohorts B and C must also resistance, or intolerance, or rejection of platinum-containing chemotherapy.

•Patients of the dose escalation phase in Part 1 must have evaluable diseases, and others must have measurable diseases as defined in RECIST V1.1 definition.

Note: The selected target lesions must meet one of two criteria: 1) no previous local treatment or 2) subsequent progression within the previous local treatment area as determined by RECIST V1.1.

* Eastern Cooperative Oncology Group (ECOG) performance status scores are 0-1.
* Expected survival is ≥3 months.
* With certain organ system functions (without transfusion, use of blood components, or G-CSF support within 14 days before testing), as defined below:

oAbsolute neutrophil count (ANC)≥1.5×10^9/L oPlatelet count (PLT)≥100×10^9/L oHemoglobin (HB)≥10 g/dL oSerum albumin≥30 g/L oTotal bilirubin≤1.5 times the upper limit of normal (ULN) oAlanine amino transferase ( ALT) and aspartate amino transferase (AST) ≤3×ULN oCreatinine≤1.5×ULN.If creatinine is>1.5×ULN, creatinine clearance is≥50 mL/min as calculated by Cockcroft-Gault formula, or urinary creatinine clearance≥50 mL/min within 24 hours as measured, the patients can still be enrolled.

* Willing and able to follow the trial and follow-up procedures.
* Capable of understanding the trial nature and voluntarily signing the written informed consent form.

Exclusion Criteria:

* Use of certain investigational drug or antineoplastic agent within 14 days or 5 half lives (whichever is longer) before first administration of investigational drug (For drugs with a longer half-life, a maximum of 4 weeks is required from the last administration; 6 weeks for chemotherapy with delayed toxicity, such as Nitroso urea or Mitomycin C).
* Execution of large surgery and radiotherapy (except focal palliative radiotherapy at least 2 weeks before first administration) within 4 weeks before first administration.
* For the dose extension stage of part 2 and part 2: having previously received systemic anti-tumor therapy exceeding three lines (excluding maintenance therapy).
* Previously received EGFR/c-Met bispecific antibody drugs (such as JNJ-61186372, EMB-01, or GB263T) for treatment.
* Prior to the first administration of the study drug, previous treatment-related toxic reactions did not alleviate to level 1 or below (CTCAE 5.0 standard), except for hair loss.
* With other malignant tumors in the past 3 years, except cancers that have been cured significantly or can be focally cured, e.g. basosquamous carcinoma of skin, carcinoma cervix in situ, or in situ breast carcinoma.
* Primary malignant tumor of the central nervous system, meningeal metastasis, or brain metastasis with spinal cord compression, or risk of cerebral hemorrhage, or symptomatic brain metastasis, or unstable brain metastasis requiring steroid and/or dehydration to reduce intracranial pressure 2 weeks before enrollment (subjects with brain metastases who are Asymptomatic or stable for more than 2 weeks after treatment and do not need steroids and/or dehydration to reduce intracranial pressure can be included in the group).
* With clinically significant cardiovascular disorder, including but not limited to:

  * Arterial thromboembolism, deep vein thrombosis or lung embolism diagnosed within 3 month before first administration of the investigational drug. Non- obstructive catheter related clot and other clinically irrelevant thrombosis are not included in the exclusion criteria. Patients with a history of related thrombosis diagnosed 3 months ago must be clinically stable for at least 4 weeks before initial administration.
  * With any of the following medical history within 6 months before first administration of the investigational drug: myocardial infarction, unstable angina, stroke, transient ischemic attack, coronary or peripheral artery bypass, or any acute coronary syndrome.
  * With abnormal ECG corrected QT interval (QTcF) at rest in the screening period. Remeasurement is made twice at intervals of more than 5 minutes. For average QTcF of 3 times ECG inspections: male: ≥ 450 msec, and female: ≥ 470 msec. With clinically significant abnormal heart rate, conduction, and ECG form at rest, e.g. complete left bundle branch block, third-degree conduction block, second-degree conduction block, and PR interval > 250 msec, double law, triple law, preexcitation syndrome, etc.
  * Poorly controlled hypertension in the investigator's opinion (systolic blood pressure > 180 mmHg, or diastolic blood pressure > 100 mmHg).
  * New York Heart Association Grade III-IV congestive heart failure, or hospitalization due to congestive heart failure within 6 months before first administration of the investigational drug.
  * Pericarditis/clinically significant pericardial effusion.
  * Cardiomyopathy.
  * ther clinically significant cardiovascular disordesr as believed by investigators.
* Active hepatitis B (hepatitis B surface antigen (HBsAg) positive and serum HBV DNA quantitative results higher than or equal to the detection limit), hepatitis C virus antibody, HIV antibody and treponema pallidum antibody positive (subjects who have a history of HCV and have completed antiviral treatment, and whose laboratory test results show that HCV-RNA is below the lower limit of quantification, can be selected for the study; those who test negative for syphilis titer can be selected).
* Patients with Interstitial lung disease, including drug-induced Interstitial lung disease or radiation pneumonia requiring long-term use of steroids or other Immunosuppressive drug in the past 1 year.
* Subjects with active gastrointestinal (GI) disease, or with a risk of GI perforation, or with other diseases that significantly interfere with the absorption, distribution, metabolism, or excretion of investigational drugs. Including but not limited to: unable to take oral medicine, uncontrollable nausea or vomiting, Bowel obstruction, inflammatory bowel disease or extensive intestinal resection, etc.
* Current severe disease or medical condition, including but not limited to uncontrolled active infection, uncontrollable pleural or abdominal effusion, and clinically significant lung, metabolic or psychiatric disorders.
* Women with child bearing potential, pregnant women or lactating women with pregnancy test positive 7 days before treatment, and male and female unwilling to take effective contraception measures or having a birth plan during the treatment and within 3 months after end of treatment.
* Subjects with a history of allergies or suspected allergic symptoms to the study drug MCLA-129, Befotertinib, or any component of both study drugs (see the investigator's brochure).
* Within one week before the first administration of the investigational drug, it is currently in use or needs to be combined with CYP3A strong inhibitors or inducers during the study period.
* Subjects still using Warfarin within 7 days before the first administration (low molecular weight heparin sodium is allowed).
* Patients poorly compliant, unable or unwilling to follow the study and/or follow-up procedures listed in the protocol, or unsuitable to participate in this trial in the investigator's opinion.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 172 (Estimated)
Dates: Start 2023-09-01 (Estimated); Primary Completion 2028-11-04 (Estimated); Study Completion 2029-07-04 (Estimated)

PRIMARY OUTCOMES:
Dose-Limiting Toxicity (DLT) | First 28 days of treatment
  To determine the dose-limiting toxicity (DLT) of MCLA-129 combined with Befotertinib in patients of advanced non-small cell lung cancer with EGFR-sensitive mutations in Part 1.
Maximum Tolerable Dose (MTD) | First 28 days of treatment
  To determine the maximum tolerated dose (MTD) of MCLA-129 combined with Befotertinib in patients of advanced non-small cell lung cancer with EGFR-sensitive mutations in Part 1.
Treatment-Emergent Adverse Event (TEAE) in Part 1 | Until 30 days after the last dosing
  To evaluate the safety of MCLA-129 combined with Befotertinib in patients of advanced non-small cell lung cancer with EGFR-sensitive mutations in Part 1 in terms of treatment-emergent adverse event (TEAE).
Overall Response Rate (ORR) in Part 2 | From date of first treatment every 6 weeks until disease progression, death or withdrawal, whichever came first, approximately 2 years
  To evaluate the efficacy of MCLA-129 combined with Befotertinib at RP2CD in patients of advanced NSCLC with EGFR-sensitive mutations in each corhort in Part 2 in terms of overall response rate (ORR)

SECONDARY OUTCOMES:
Overall Response Rate (ORR) in Part 1 | From date of first treatment every 6 weeks until disease progression, death or withdrawal, whichever came first, approximately 2 years
  To evaluate the efficacy of MCLA-129 combined with Befotertinib at RP2CD in patients of advanced NSCLC with EGFR-sensitive mutations in each corhort in Part 1 in terms of overall response rate (ORR).
Disease Control Rate (DCR) in Part 1 and 2 | From date of first treatment every 6 weeks until disease progression, death or withdrawal, whichever came first, approximately 2 years
  To evaluate the efficacy of MCLA-129 combined with Befotertinib at RP2CD in patients of advanced NSCLC with EGFR-sensitive mutations in patients with advanced NSCLC and other solid tumors in Part 1 and 2 in terms of disease control rate (DCR).
Progression-Free Survival (PFS) in Part 1 and 2 | From date of first treatment every 6 weeks until disease progression, death or withdrawal, whichever came first, approximately 2 years
  To evaluate the efficacy of MCLA-129 combined with Befotertinib at RP2CD in patients of advanced NSCLC with EGFR-sensitive mutations in patients with advanced NSCLC and other solid tumors in Part 1 and 2 in terms of Progression-free survival (PFS).
Duration of Response (DOR) in Part 1 and 2 | From date of first treatment every 6 weeks until disease progression, death or withdrawal, whichever came first, approximately 2 years
  To evaluate the efficacy of MCLA-129 combined with Befotertinib at RP2CD in patients of advanced NSCLC with EGFR-sensitive mutations in patients with advanced NSCLC and other solid tumors in Part 1 and 2 in terms of duration of response (DOR).
Anti-Drug Antibody (ADA) in Part 1 and 2 | Until 30 days after the last dosing
  To assess the Incidence of anti-drug antibodies in serum blood against MCLA-129 following administration of MCLA-129.
Overall Survival (OS) in Part 2 | From date of first treatment every 6 weeks until death or withdrawal, whichever came first, approximately 2 years
  To evaluate the efficacy of MCLA-129 combined with Befotertinib at RP2CD in patients of advanced NSCLC with EGFR-sensitive mutations in Part 2 in terms of overall survival (OS).
Treatment-Emergent Adverse Event (TEAE) in and 2 | Until 30 days after the last dosing
  To evaluate the safety of MCLA-129 combined with Befotertinib in patients of advanced non-small cell lung cancer with EGFR-sensitive mutations in Part 2 in terms of treatment-emergent adverse event (TEAE).
Maximum plasma concentration [Cmax] | Until 30 days after the last dosing
  To evaluate the PK profile of MCLA-129 combined with Befotertinib in patients dvanced NSCLC with EGFR-sensitive mutations in Part 1.
Time to reach maximum concentration [Tmax] | Until 30 days after the last dosing
  To evaluate the PK profile of MCLA-129 combined with Befotertinib in patients dvanced NSCLC with EGFR-sensitive mutations in Part 1.
Trough concentration [Ctrough] | Until 30 days after the last dosing
  To evaluate the PK profile of MCLA-129 combined with Befotertinib in patients dvanced NSCLC with EGFR-sensitive mutations in Part 1.
Area under the concentration [AUC] | Until 30 days after the last dosing
  To evaluate the PK profile of MCLA-129 combined with Befotertinib in patients dvanced NSCLC with EGFR-sensitive mutations in Part 1.

CONTACTS AND LOCATIONS:
Overall Officials: Shun Lu, M.D., Study Chair — Shanghai Chest Hospital
Locations (3):
- China (3):
  - The first affiliated hospital of bengbu medical college, Bengbu, Anhui
  - Hunan cancer hospital, Changsha, Hunan
  - Shanghai chest hospital, Shanghai

IPD SHARING:
Plan to Share IPD: No